CLINICAL TRIAL: NCT06135142
Title: Comparison Of The Effects Of Connective Tissue Massage And Classical Massage On Pain, Functional Status And Quality Of Life In Patients With Chronic Non-Specific Low Back Pain.
Brief Title: Connective Tissue Massage And Classical Massage In Patients With Chronic Non-Specific Low Back Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cansu DAL (Other)
Responsible Party: Sponsor-Investigator, Cansu DAL, Principal Investigator, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CD1
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Connective Tissue Massage; Classical Massage; Lumbar Mobility; Quality of Life
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation; Diathermy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Connective Tissue Massage Group (Experimental): The patient was positioned in sitting position and their feet were supported.The basic region consisted of short and long strokes to the anterior superior iliac spine, the sacrolumbar angle, the ilium, L5 to T12, the pectoral muscles.After,the transition was made to the lower thoracic region.Short strokes were applied from lateral to medial on the latissimus dorsi muscle.Short strokes were executed between the transverse processes of the vertebrae from T12 to T7.Following this,long strokes were initiated from the axilla and continued up to the vertebrae.Finally,long strokes continued beneath the scapular angles.At the end of the lower thoracic region massage,the pectoral muscles were subjected to three stroking motions.After concluding the massage of the lower thoracic region,the application was finalized with long strokes performed subcostally and under the iliac crest.
  Interventions: Other: Connective Tissue Massage
- Classic Massage Group (Experimental): The patient positioned themselves face down with their upper clothing removed. The massage initiation involved employing a general stroking motion. Commencing from the sacrolumbar region, paravertebral long sweeping strokes were executed bilaterally, progressing upwards along the vertebrae's lateral edges. In the area spanning from the lumbothoracic boundary to the gluteals, a general stroking motion was iterated thrice. Subsequently, the erector spinae, latissimus dorsi, and gluteus maximus muscles were sequentially subjected to a series of actions: three cycles of stroking, followed by three cycles of kneading, concluding with three more cycles of stroking. As a concluding step, the initial general stroking movements were replicated thrice prior to finalizing the massage session.
  Interventions: Other: Classical Massage
- Control Group (Active Comparator): The standardized physiotherapy program included the application of superficial thermal heat, transcutaneous electrical nerve stimulation (TENS) and therapatic Ultrasound. TENS at a frequency of 100 Hz (250-μsec pulses) was applied for 15 min using two 4- to 6-cm electrodes placed bilaterally on each side of the spinous process of the L4 to S1 vertebrae with thermal therapy. While the TENS application was in progress, the heat treatment was also applied. Topical moist heat treatment at 40°C applied directly on the skin to increase both tissue temperature and blood flow. Then, continuous ultrasound was applied at an intensity of 1.5 to 2.5 W/cm2 for a period of 5 minutes.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Device: Therapatic Ultrasound; Other: Heat Treatment

INTERVENTIONS:
Other: Connective Tissue Massage — It involves manipulating the soft and deep tissues of the body.
  Arms: Connective Tissue Massage Group
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — The sum of therapeutic modalities of physical medicine capable to change the threshold of elicitation of nerve or muscle.
  Arms: Control Group
Other: Classical Massage — It involves manipulating the soft tissues of the body.
  Arms: Classic Massage Group
Device: Therapatic Ultrasound — The sum of therapeutic modalities of physical medicine capable to change the threshold of elicitation of nerve or muscle.
  Arms: Control Group
Other: Heat Treatment — Applying heat to an affected area to treat damaged muscles, joints or tissues in the body.
  Arms: Control Group

SUMMARY:
Objective This study aimed to compare the effects of connective tissue massage and classical massage on pain, functional status and quality of life in patients with chronic non-specific low back pain.

Methods The study included 30 participants diagnosed with chronic non-specific low back pain. Participants were randomly divided into three groups: classical massage (n=10), connective tissue massage (n=10), and control groups (n=10). The control group received standart physical therapy only. All interventions were administered over a period of 3 days per week for 4 weeks, with each session lasting approximately 15-20 minutes. All assessments were performed at baseline and at the end of 4 weeks. For all participants, the severity of pain was assessed using the Visual Analog Scale, the level of impaired function was measured using the Functional Low Back Pain Scale, lumbar mobility was evaluated with the Modified Schober Test and Sit and Reach Test, physical disabilities were gauged using the Roland Morris Disability Questionnaire, and the quality of life was assessed using the Short Form-36 Quality of Life questionnaire.

DETAILED DESCRIPTION:
This was a 3-arm randomized controlled trial, parallel-group study with blind outcomes assessor. Ethical approval was obtained from the Muğla Sıtkı Koçman University Health Sciences Ethics Committee (09.01.2020, decision no: 4). Detailed information about the study was verbally provided to participants, and written informed consent was obtained. The study adhered to the ethical principles of the Helsinki Declaration. The study design adhered to the CONSORT guidelines for rigorous reporting.11 After obtaining consent and confirming the inclusion criteria, a convenience sample of 30 participants was equally and randomly divided into three groups: the CTM group (n=10), CM group (n=10), and control group (n=10). Randomization was carried out by an independent physical therapist, who was not involved in the assessment or treatment of the participants, 1 hour before the baseline measurements. The randomization process involved using opaque and sealed envelopes, each containing a group allocation number generated from a computer-generated random number table. Block randomization was employed to ensure an equal distribution of participants across the groups.

All treatment sessions were administered by the same investigator (C.D) in the study group. The intervention duration was uniform across all groups: 4 consecutive weeks, with 3 sessions per week lasting 15-20 minutes per session. Outcome measurements were taken at the beginning and 4 weeks after the completion of the program. An independent physiotherapist, unaware of the research details and participant groupings, conducted the evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65,
* Diagnosis of chronic non-specific low back pain,
* Rest or activity pain score of 3 or higher on the Visual Analog Scale (VAS).

Exclusion Criteria:

* Undergoing surgical operation within the last 6 months or having prior spinal surgery,
* Presence of spondyloarthropathy, spondylolisthesis, or lumbar stenosis,
* Systemic inflammatory disease,
* Usage of non-specific anti-inflammatory medication in the past 15 days
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-12-08 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 weeks
  The VAS is a widely used, valid, and reliable measurement method for assessing pain intensity. It consists of a horizontal line drawn to a length of 10 cm, with the numbers 0 and 10 located at the left and right ends, respectively. Zero represents "no pain at all," while 10 represents "the most severe pain imaginable." As one moves from left to right along the line, the intensity of pain increases. The patient is asked to mark on the VAS where their current pain intensity lies, based on how they feel at the moment of assessment. The measurement is then recorded in centimeters using a ruler .
Modified Schober Test (MST) | 4 weeks
  The MST is used to assess lumbar mobility in patients. Two Spina iliaca posterior superior landmarks are identified and connected by drawing a line to mark the midline. A point is marked 10 cm above and 5 cm below this midline. The distance between these two points should be 15 centimeters. Subsequently, the patient is asked to bend forward from the waist without bending the knees. While bending, the distance between the same two points is measured again, and the amount of change is calculated.
Sit and Reach Test (SRT) | 4 weeks
  The SRT, can be utilized to assess trunk mobility or flexibility in patients with back pain. The test was performed by sit and reach box with a measuring scale. The test involved sitting on the floor with legs stretched out straight ahead. The soles of the feet were placed flat against the box. Both knees were locked and pressed flat to the floor. With the palms facing downward and the hands on top of each other, the subjects reached forward along the measuring line as far as possible. The points reached by the patients were marked and recorded.
Back Pain Functional Scale (BPFS) | 4 weeks
  The BPFS is a 12-item scale used to assess how patients' activities and functions are affected by their current back pain complaints. The scale evaluates activities related to work, school, household tasks, general habits, forward bending, putting on shoes/socks, lifting objects from the ground, sleeping, sitting, standing, walking, stair climbing, and driving a car. For patients who do not drive, the final question can be answered as "travelling." Each statement is scored from 0 to 5, with a maximum score of 60 and a minimum score of 0. Higher scores indicate less difficulty in performing functional activities.
Roland Morris Disability Qustionnaire (RMDQ) | 4 weeks
  The RMDQ, is a patient-administered scale consisting of 24 items used to assess patients' functional status.Patients are asked to respond to statements that correspond to their current condition, leaving blank spaces for statements that do not apply to them. Each answered statement is assigned a score of 1, and the total score of the questionnaire is calculated. The change in the total questionnaire score is used to determine the clinical improvement rate.
Short Form-36 Questionnaire (SF-36) | 4 weeks
  The SF-36 is a patient-administered questionnaire consisting of 36 items used to assess an individual's quality of life. It includes two sections, namely physical health (physical functioning, physical role, pain, general health) and mental health (vitality, social functioning, emotional role, mental health), with a total of eight subdomains. Each subdomain is scored on a scale of 0 to 100. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Cansu DAL, Principal Investigator — Muğla Sıtkı Koçman University; Meltem KOÇ, Study Director — Muğla Sıtkı Koçman University; Banu BAYAR, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Bayındır Devlet Hastanesi, Izmir, Bayındır, Turkey (Türkiye)